CLINICAL TRIAL: NCT06347601
Title: Survey on Sexual Harassment and Gender Discrimination in the Healthcare Sector in Taiwan
Brief Title: Survey on Sexual and Gender in the Healthcare in Taiwan
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-03-011AC
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sexual Harassment
MeSH Terms: conditions — Sexual Harassment | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Without Intervention — Without Intervention

SUMMARY:
This study addresses the pervasive issue of sexual harassment within Taiwanese society, particularly within the medical field, where comprehensive research is lacking. The research objective is to explore patterns of sexual harassment and gender discrimination experiences among physicians and medical students in Taiwan, while also investigating potential associations with professional burnout and mental health. Employing a convergent mixed-methods design, the study combines quantitative surveys and qualitative in-depth interviews. While lacking a control group and utilizing non-blinding methods without random assignment, the study aims to recruit 1000 participants aged 18 or older, considering both valid responses and potential dropouts. Additionally, interviews will be conducted with 30 individuals who have experienced sexual harassment or are interested in gender issues. The research methods will assess sexual harassment experiences, professional burnout, and depressive symptoms as primary outcomes or indicators.

ELIGIBILITY:
Inclusion Criteria:

Taiwanese medical students or physicians Aged 18 or older Have received education or practiced in Taiwan's medical colleges or hospitals

Exclusion Criteria:

Individuals under 18 years old Have not received education or practiced in Taiwanese medical colleges or hospitals Unable to understand or complete Chinese-language questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes Taiwanese medical students and physicians who meet the following criteria:
  Inclusion Criteria:
  Aged 18 years or older. Have received education or practiced in Taiwan's medical colleges or hospitals. Voluntarily agree to participate in the research through questionnaire surveys or interviews.
  Exclusion Criteria:
  Individuals under 18 years old. Those who have not received education or practiced in Taiwanese medical colleges or hospitals.
  Those unable to understand or complete Chinese-language questionnaires. Those unable to participate in interviews.
Sampling Method: Non-Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | One year
  Center for Epidemiologic Studies Depression Scale consists of 20 items. The total score can range from 0 to 60. Higher scores indicate greater depressive symptoms. Lower scores suggest fewer depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No